CLINICAL TRIAL: NCT06441708
Title: Neutrophil Extracellular Traps (NETs) Mediated Killing of Carbapenem-resistant Pseudomonas Aeruginosa Isolated From Hospital Acquired Infections in Assiut University Hospitals
Brief Title: Neutrophil Extracellular Traps (NETs) Mediated Killing of Carbapenem-resistant Pseudomonas Aeruginosa.
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, NSHussein, Assistant Lecturer at medical Microbilogy and Immunology department, Assiut University
Other Study IDs: Pseudomonas aeruginosa
Record Dates: First submitted 2024-05-29; First posted 2024-06-04 (Actual); Last update posted 2024-06-04 (Actual); Status verified 2024-06

CONDITIONS: Neutrophil Extracellular Traps Formation

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: No intervention — No intervention on patient

SUMMARY:
Aim of the work:

To determine the killing ability of neutrophils to ATCC 27853, carbapenem-resistant P. aeruginosa.

To compare between the ability of ATCC 27853, carbapenem-resistant P. aeruginosa to induce NETs formation.

To quantify NETS formation in response to PMA, ATCC 27853, carbapenem-resistant P. aeruginosa using immunofluorescence.

To determine the killing ability of NETs on ATCC 27853, carbapenem-resistant P. aeruginosa.

DETAILED DESCRIPTION:
Pseudomonas aeruginosa is one of the most common pathogens in healthcare-associated infections worldwide, causing ventilator-associated pneumonia, urinary tract infections in patients with long-term urinary catheterization, wound infections, bloodstream infections, and otitis (reynolds and kollef, 2021).

Carbapenem-resistant-P. aeruginosa infection is a prominent disease connected to healthcare due to multiple mechanisms, such as target alteration, active efflux, decreased permeability, and enzyme degradation (Tenover et al., 2022).

Neutrophils are the most prominent cellular component of the innate immune response and are essential for defense against bacterial infections (Chapple et al., 2023).

In addition to traditional antimicrobial processes of neutrophils, a unique web-like structure, is termed neutrophil extracellular traps (NETs), formed and released by highly active neutrophils. NETs consist of extracellular deoxyribonucleic acid (eDNA) filaments coated with histones and neutrophil granule proteins such as Myeloperoxidase (MPO), neutrophil elastase (NE), lactoferrin, cathepsins, calprotectin, LL-37, and defensin (Papayannopoulos, 2018).

MPO and NE are key components of NETs and play roles in their function and structure. MPO, a heme protein primarily stored in the granules of neutrophils, contributes significantly to microbial killing within NETs. It catalyzes the production of hypochlorous acid from hydrogen peroxide and chloride ions, a reaction central to the antimicrobial properties of NETs. NE, another granule protein extends to modulating inflammation and immune response (Islam et al., 2023).

The role of NETs during bacterial infection is not completely clear. It promoted the clearance of bacteria by facilitating the entrapping and killing of these pathogens, However, it has been described that the granular proteins released within the NETs act mainly as a regulator of inflammation due to the action on different cytokines, rather than as a bactericidal mechanism (Clancy, 2018).

P. aeruginosa-mediated factors contribute to the NETosis and release of a large amount of NETs. However, sequestration of P. aeruginosa by traps does not lead to the complete destruction of bacteria, but, it promotes their microcolonization, aggregation, and finally biofilm formation, leading to the formation of higher resistance to NETs-mediated bactericidal activity (Rahman and Gadjeva, 2014).

Neutrophils formed a NET-barrier to keep bacteria outside in the form of biofilm and prevent their spread to the brain. Thus, the NET formation is probably a useful mechanism for protecting the brain against infections through the ocular route (Thanabalasuriar et al., 2019).

ELIGIBILITY:
Inclusion Criteria:

* isolates will be isolated from different clinical samples including wound respiratory tract urine and blood. _carbapenem-resistant P. aeruginosa isolates.

Exclusion Criteria:

* _carbapenem-sensitive P. aeruginosa isolates.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Clinical isolates from different clinical samples including urine, blood, sputum, wound
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2024-06-01 (Estimated); Primary Completion 2025-06-01 (Estimated); Study Completion 2025-07-01 (Estimated)

PRIMARY OUTCOMES:
Quantitification of neutrophils extracellular traps by immunofluroscrnce | Three months
  Quantitification of neutrophils extracellular traps by indirect immunofluroscrnce